CLINICAL TRIAL: NCT00134277
Title: Prospective Randomised Comparing Trial Between an Infragenual Dilatation (ID), an ID With Stenting, an ID With Cutting Balloon and Laser Therapy
Brief Title: Trial Comparing Different Medical Devices for Infragenual Dilatation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/161
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Diabetic Angiopathies; Intermittent Claudication
MeSH Terms: conditions — Diabetic Angiopathies; Intermittent Claudication | interventions — Stents; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Infragenual dilatation with stenting (Active Comparator)
  Interventions: Procedure: Infragenual dilatation with stenting
- Infragenual dilatation with cutting balloon (Active Comparator)
  Interventions: Procedure: Infragenual dilatation with cutting balloon
- Laser therapy (Active Comparator)
  Interventions: Procedure: Laser therapy
- Infragenual dilatation (Placebo Comparator)
  Interventions: Procedure: Infragenual dilatation

INTERVENTIONS:
Procedure: Infragenual dilatation — Infragenual dilatation
  Arms: Infragenual dilatation
Procedure: Infragenual dilatation with stenting — Infragenual dilatation with stenting
  Arms: Infragenual dilatation with stenting
Procedure: Infragenual dilatation with cutting balloon — Infragenual dilatation with cutting balloon
  Arms: Infragenual dilatation with cutting balloon
Procedure: Laser therapy — Laser therapy
  Arms: Laser therapy

SUMMARY:
This study is a comparison of different medical devices for infragenual dilatation.

DETAILED DESCRIPTION:
Dilatation and recanalisation of the distal veins (infragenual popliteal artery, tibiofibular trunc, posterior tibial artery, anterior tibial artery) by classical balloon dilatation or cutting balloon with or without stenting or by endovascular laser. This intervention happens only once; the duration of the intervention depends on the procedure and the original injuries(30 - 120 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type I or II with diabetic angiopathy stage IIb to IV (Fontaine)
* Atherosclerotic patients with distal angiopathy stage IIb to IV (Fontaine)

Exclusion Criteria:

* Acute ischemia
* Multisegmentaric damage above the knee
* Sepsis: acute respiratory distress syndrome (ARDS), C-reactive protein (CRP) > 30, white blood cell (WBC) > 25,000
* Acute myocardial infarction (AMI) during the last 14 days
* Operative contraindication
* Life expectancy < 2 years
* Blue toe syndrome (micro-embolisation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-09; Primary Completion 2009-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Primary patency after 6 months | After 6 months

SECONDARY OUTCOMES:
Proving the superiority or non-superiority of one treatment procedure to another treatment procedure | After 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Caren Randon, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be